CLINICAL TRIAL: NCT03489473
Title: FESPET Study: Female EStrogen recePtor in Endometrial Cancer Treatment
Acronym: FESPET
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); University Medical Center Groningen (Other); Haukeland University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: FESPET
Record Dates: First submitted 2018-03-12; First posted 2018-04-05 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-03

CONDITIONS: Endometrial Cancer
Keywords: Hormonal therapy; FES PET scan; Estrogen receptor
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: 18F-FES PET CT scan — PET CT scan with estrogen tracer

SUMMARY:
Endometrial cancer is the most common gynecological malignancy in the western world and its incidence is expected to increase in the coming years due to obesity. Major treatment modalities include surgery, radiotherapy and chemotherapy. Hormonal therapy can be considered in primary treatment if other treatment modalities are not feasible and in treatment for recurrent disease. Hormonal treatment has shown to be more effective in endometrial cancers expressing estrogen (ER) and progesterone receptor (PR). Tumor heterogeneity frequently causes loss of expression of ER and PR in metastasis compared to primary tumors. The FES PET CT scan combines PET-CT scan with an estrogen tracer, thus allowing non invasive visualisation of estrogen receptor, even in patients with metastasis that are difficult to reach for biopsy. FES PET has been shown to relate well to ER expression and to treatment response in breast cancer. This study explores the feasibility of the FES PET scan in endometrial cancer patients.

DETAILED DESCRIPTION:
Endometrial carcinoma is the most common gynecological malignancy in the western world, and with a current incidence of 18/100.000 women per year in the European Union, it affects around 65,000 new women each year. Due to the increased life expectancy and obesity, the incidence of endometrial cancer has increased in the last years, and is expected to rise in the coming years. Most patients present with early stage disease and have a favorable outcome. However, patients with metastatic disease have few treatment options with a poor prognosis.

Surgery is the primary treatment modality in endometrial cancer and defines the final surgicopathological stage according to the International Federation of Gynecology and Obstetrics (FIGO) staging system. Adjuvant treatment is based on final tumor grade and FIGO stage and consists of radiotherapy and-or chemotherapy. Hormonal therapy is considered as alternative treatment modality for: 1. patients who are not suitable for surgery, 2. patients who wish to maintain fertility, and 3. patients with metastatic disease. A recent review summarizes the available evidence on the effect of hormonal therapy in patients with advanced and recurrent endometrial cancer. The overall response rate based on a single biopsy taken prior to treatment, was 22%. In ER positive tumors, the response rate was 27% compared to 9% in ER negative tumors. In PR positive tumors 36% of patients responded, compared to 12% in PR negative tumors. Thus, the presence of ER and PR receptors on the tumor cell seems to be relevant for prediction of response to hormonal treatment. Yet, data concerning the percentage of ER and PR expression are lacking, and might underestimate the response to hormonal treatment in individual cases.

Analysis of the genomic landscape of endometrial cancer has shown marked genetic heterogeneity between biopsies of primary tumors and their corresponding metastases, suggesting that only a part of tumor cells in the primary tumor is involved in metastases. Also, loss of ER and PR expression is frequently observed in metastases from ER/PR positive primary tumors. These findings underline the relevance of obtaining a new biopsy to determine ER and PR expression in recurrent disease. This can be challenging since recurrences can be hard to reach by biopsies due to its location and multiplicity.

18F-FES PET CT (FES PET) is a novel imaging method based on positron emission tomography using a specific tracer targeting ER allowing the visualization of ER expression in tissue. FES PET allows non-invasive depiction and quantification of ER expression in all tumor lesions in a patient.

FES PET has been evaluated in breast cancer with a reported sensitivity of 69% to 100%, and a specificity of 80-100% for identifying ER positive tumor when compared to immunohistochemical expression of ER. In endometrial cancer, FES PET has been evaluated in only two studies. The first study included 19 patients with endometrial cancer with different FIGO stages that underwent FES PET prior to surgical resection. In this study a significant correlation between ER uptake on FES PET and ER immunohistochemical expression was observed. In the second study 22 patients were analyzed and classified into high risk (FIGO stage ≥Ic or grade ≥2) and low risk (FIGO stage ≤1b and grade 1) endometrioid type endometrial carcinoma. In the high risk group a significantly lower FES uptake was observed when compared to the low risk group, suggesting that FES PET could assist in identifying patients with high risk endometrial cancer. As shown by van Kruchten et al., FES PET could also be of value in the evaluation of response to hormonal therapy. In this study the results of serial FES PET scans are described in 16 patients with metastatic breast cancer treated with fulvestrant, a selective estrogen downregulator. Response to hormonal therapy was associated with reduced uptake on subsequent FES PET scans. So far, FES PET data are limited in endometrial cancer to one case report in which a decrease of estrogen uptake was observed upon medroxyprogesterone therapy in early stage endometrial cancer consistent with histological and clinical follow-up. Based on previous findings the aim of the current study is to explore the feasibility of FES PET scan in patients with endometrial cancer.

ELIGIBILITY:
Inclusion Criteria:

* Primary or metastatic endometrial cancer in which hormonal treatment is the planned treatment
* Postmenopausal status
* All histologic types of endometrial cancer (e.g. endometrioid, clear cell, serous subtype)
* Availability of recent (micro)curettage or biopsy

Exclusion Criteria:

* Intercurrent treatment between biopsy taking and start of hormonal treatment
* Sarcoma of the uterus
* Contra-indications to perform a PET-CT scan or a CT scan with intravenous contrast
* Use of hormonal therapy in the three months preceding performance of FES PET

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Gender identity since the study population is found in patients with endometrial cancer
Study Population: Patient with either
  * Primary endometrial cancer and planned hormonal treatment
  * Recurrent endometrial cancer and planned hormonal treatment
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
estrogen uptake on FES PET scan | Within 1 month of inclusion
  Standard uptake volume of FES

SECONDARY OUTCOMES:
Estrogen and Progesterone Receptor expression | Within 1 month of inclusion
  Percentage of tumor cells expressing estrogen and progesterone receptor through immunohistochemical analysis of tissue biopsy material

CONTACTS AND LOCATIONS:
Overall Officials: JMA Pijnenborg, MD, PhD, Principal Investigator — Radboud University Medical Center

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers. This will be decided when a request for sharing of IPD is made

REFERENCES:
- [Background] Basen-Engquist K, Chang M. Obesity and cancer risk: recent review and evidence. Curr Oncol Rep. 2011 Feb;13(1):71-6. doi: 10.1007/s11912-010-0139-7. PMID 21080117
- [Background] Carlson MJ, Thiel KW, Leslie KK. Past, present, and future of hormonal therapy in recurrent endometrial cancer. Int J Womens Health. 2014 May 2;6:429-35. doi: 10.2147/IJWH.S40942. eCollection 2014. PMID 24833920
- [Background] Amant F, Mirza MR, Koskas M, Creutzberg CL. Cancer of the corpus uteri. Int J Gynaecol Obstet. 2015 Oct;131 Suppl 2:S96-104. doi: 10.1016/j.ijgo.2015.06.005. No abstract available. PMID 26433681
- [Background] Ethier JL, Desautels DN, Amir E, MacKay H. Is hormonal therapy effective in advanced endometrial cancer? A systematic review and meta-analysis. Gynecol Oncol. 2017 Oct;147(1):158-166. doi: 10.1016/j.ygyno.2017.07.002. Epub 2017 Jul 6. PMID 28689667
- [Background] Gibson WJ, Hoivik EA, Halle MK, Taylor-Weiner A, Cherniack AD, Berg A, Holst F, Zack TI, Werner HM, Staby KM, Rosenberg M, Stefansson IM, Kusonmano K, Chevalier A, Mauland KK, Trovik J, Krakstad C, Giannakis M, Hodis E, Woie K, Bjorge L, Vintermyr OK, Wala JA, Lawrence MS, Getz G, Carter SL, Beroukhim R, Salvesen HB. The genomic landscape and evolution of endometrial carcinoma progression and abdominopelvic metastasis. Nat Genet. 2016 Aug;48(8):848-55. doi: 10.1038/ng.3602. Epub 2016 Jun 27. PMID 27348297
- [Background] Geels YP, van der Putten LJM, van Tilborg AAG, Nienhaus BEC, van den Berg-van Erp SH, Snijders MPLM, van der Wurff A, Massuger LFAG, Bulten J, Pijnenborg JMA. Immunohistochemical Profiles of Endometrioid Endometrial Carcinomas With and Without Metastatic Disease. Appl Immunohistochem Mol Morphol. 2018 Mar;26(3):173-179. doi: 10.1097/PAI.0000000000000402. PMID 27299188
- [Background] Vandenput I, Trovik J, Leunen K, Wik E, Stefansson I, Akslen L, Moerman P, Vergote I, Salvesen H, Amant F. Evolution in endometrial cancer: evidence from an immunohistochemical study. Int J Gynecol Cancer. 2011 Feb;21(2):316-22. doi: 10.1097/IGC.0b013e31820575f5. PMID 21734474
- [Background] Tsujikawa T, Yoshida Y, Kiyono Y, Kurokawa T, Kudo T, Fujibayashi Y, Kotsuji F, Okazawa H. Functional oestrogen receptor alpha imaging in endometrial carcinoma using 16alpha-[(1)(8)F]fluoro-17beta-oestradiol PET. Eur J Nucl Med Mol Imaging. 2011 Jan;38(1):37-45. doi: 10.1007/s00259-010-1589-8. Epub 2010 Aug 18. PMID 20717823
- [Background] Tsujikawa T, Yoshida Y, Kudo T, Kiyono Y, Kurokawa T, Kobayashi M, Tsuchida T, Fujibayashi Y, Kotsuji F, Okazawa H. Functional images reflect aggressiveness of endometrial carcinoma: estrogen receptor expression combined with 18F-FDG PET. J Nucl Med. 2009 Oct;50(10):1598-604. doi: 10.2967/jnumed.108.060145. Epub 2009 Sep 16. PMID 19759112
- [Background] van Kruchten M, de Vries EG, Glaudemans AW, van Lanschot MC, van Faassen M, Kema IP, Brown M, Schroder CP, de Vries EF, Hospers GA. Measuring residual estrogen receptor availability during fulvestrant therapy in patients with metastatic breast cancer. Cancer Discov. 2015 Jan;5(1):72-81. doi: 10.1158/2159-8290.CD-14-0697. Epub 2014 Nov 7. PMID 25380844
- [Background] Yoshida Y, Kurokawa T, Sawamura Y, Shinagawa A, Okazawa H, Fujibayashi Y, Kotsuji F. The positron emission tomography with F18 17beta-estradiol has the potential to benefit diagnosis and treatment of endometrial cancer. Gynecol Oncol. 2007 Mar;104(3):764-6. doi: 10.1016/j.ygyno.2006.10.024. Epub 2006 Dec 6. PMID 17156828
- [Background] Trovik J, Wik E, Werner HM, Krakstad C, Helland H, Vandenput I, Njolstad TS, Stefansson IM, Marcickiewicz J, Tingulstad S, Staff AC; MoMaTEC study group; Amant F, Akslen LA, Salvesen HB. Hormone receptor loss in endometrial carcinoma curettage predicts lymph node metastasis and poor outcome in prospective multicentre trial. Eur J Cancer. 2013 Nov;49(16):3431-41. doi: 10.1016/j.ejca.2013.06.016. Epub 2013 Aug 8. PMID 23932335
- [Background] Tangen IL, Werner HM, Berg A, Halle MK, Kusonmano K, Trovik J, Hoivik EA, Mills GB, Krakstad C, Salvesen HB. Loss of progesterone receptor links to high proliferation and increases from primary to metastatic endometrial cancer lesions. Eur J Cancer. 2014 Nov;50(17):3003-10. doi: 10.1016/j.ejca.2014.09.003. Epub 2014 Sep 30. PMID 25281525
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774